CLINICAL TRIAL: NCT03773627
Title: MRI Marker of Postoperative Delirium and Delayed Neurocognitive Recovery
Brief Title: MRI Maker of Perioperative Neurocognitive Disorder
Acronym: MRIPND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-075
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Necrosis of Femoral Head; Knee Osteoarthritis; Fracture of Lower Limb
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Periperative neurocognitive disorder(PND) is consistently associated with increased morbidity and mortality, but its mechanisms remain unclear. Moreover, valid biomarkers for the prediction or diagnosis of the development of delayed neurocognitive recovery in aged patients have not been identified so far. The purpose of this study is trying to find the functional MRI marker of PND.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* Spoke proficient Chinese
* Selected to lower limb osteopathic surgery
* Informed consent signed by the patient
* Underwent general anesthesia

Exclusion Criteria:

* Existing cerebral disease, or have a history of neurological and psychiatric diseases including AD, stroke, and psychosis
* Existing cognitive impairment as evidenced by Mini-Mental State Examination scores below 24
* Several audition or vision disorder
* With standard contraindications to MRI examinations
* Unwillingness to comply with the protocol or procedures.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients elder than 60 years old elective to undergo lower limb surgery and conform to the including criteria would be recruited.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-12-12 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
MRI markers of PND before 7th day after surgery | From the day before surgery to the 7th day after surgery
  To analysis the association of volume of hippocampus measured by MRI and the occurrence of PND identified at the 7th day after surgery

SECONDARY OUTCOMES:
MRI markers of PND before 12 month after surgery | From the 7th day after surgery to 12 month after surgery
  To analysis the association of volume of hippocampus measured by MRI and the occurrence of PND identified at the 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: qi lu, Dr., Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided